CLINICAL TRIAL: NCT02232126
Title: Social Work Intervention Focused on Transitions Among At-Risk Older Adults
Brief Title: Social Work Intervention Focused on Transitions
Acronym: SWIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Huntington Hospital (Other Government); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Susan Enguidanos, Associate Professor of Gerontology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: UP-10-00372; 5R21AG034557-02 (NIH)
Record Dates: First submitted 2014-08-25; First posted 2014-09-05 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Study Focus: 30-day Rehospitalizations Among At-risk Older Adults Randomized to a Social Work-driven Care Transitions Intervention; Heart Disease; Diabetes; Hypertension; Cancer; Depression; Asthma; Chronic Heart Failure; Chronic Obstructive Pulmonary Disease; Stroke
Keywords: Hospital readmissions; Randomized controlled trial; Older adults; Care transitions; Social work
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus; Hypertension; Neoplasms; Depression; Asthma; Pulmonary Disease, Chronic Obstructive; Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention)
- Intervention (Experimental)
  Interventions: Other: SWIFT home intervention

INTERVENTIONS:
Other: SWIFT home intervention — 1 in-home assessment performed by study social worker, another in-home visit performed if needed. Up to 4 telephone contacts performed by study social worker. A maximum of 6 contacts
  Arms: Intervention

SUMMARY:
In response to Program Announcement (PA)-09-164, "NIH Exploratory/Developmental Research Grant Program (R21) a randomized pilot study testing the efficacy of SWIFT: Social Work Intervention Focused on Transitions among at-risk older adults following hospital discharge to home. This study is drawn from several observations. First, transitions between care settings create elevated risk for poor outcomes and for readmission among older adults leaving the hospital for home largely due to fragmented care and poor communication. Next, while few studies exist that test methods to improve transitions, those available are largely medically focused, using a nurse or advanced practice nurse in their approach. Although evidence exists to support the effectiveness of these models, few have been replicated and none have been integrated into standard health care practice. This may be attributed to several factors including the availability of the needed staff, the lack of existing structures to support these roles, and the costs of implementing these interventions. Finally, a social work driven intervention may provide a replicable mechanism for bridging medical care, addressing psychosocial needs as well as medical needs, and improving linkages with community services while reducing care duplication. This study aimed to test a structured social work transition intervention model to reduce rates of hospital readmission and medical service use while improving patient satisfaction with the care transition process. A randomized pilot study was used to test a social work transitions model designed to improve care provided to frail older adults being discharged from the hospital to return to the community. Eligible patients consenting to participate (n=181) were randomly assigned to either the social work transitions model intervention or usual care. This project was conducted at Huntington Hospital, a 525-bed, nonprofit, community hospital located in Pasadena, California. In an average year, Huntington Hospital has approximately 10,000 older adults discharged from their facility, 44% of who are 80 years old or older. Those randomized to the intervention arm received up to six sessions from the social worker, at least one provided in the home. The social work intervention was designed to overcome common problems following hospital discharge including medication review, discussion and planning around discharge instruction, assistance in scheduling follow up appointments, assessments of psychosocial and other support service needs and provision of linkages to address those needs. Outcomes were measured three and six months following arrival at home, with an interim measure of satisfaction at 10 days following arrival at home, with measures including patient level of depression, pain, physical functioning, self-efficacy with disease management, and medical service use.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or more
* English-speaking
* Community dwelling (own home, vs. assisted living facility/skilled care)
* Living within specified service net
* Cognitively intact (as measured by a score of 5 or more on the SPMSQ)
* Meeting at lease one or more of the following:
* Age 75 or more
* Taking 5 or more prescription medications
* Had at least one inpatient admission or emergency department visit in previous 6 months

Exclusion Criteria:

* Age 64 or younger
* Non-English speaking
* Diagnosed with end-stage renal disease
* Hospice recipient
* Diagnosis of Alzheimer's disease or severe dementia
* Residing in assisted living or skilled care facility
* Homeless

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 181 (Actual)
Dates: Start 2011-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Huntington Hospital, Pasadena, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 91 | 90
Completed | 91 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Usual care consisted of the usual course of care provided to older adults transitioning home from a hospital stay at Huntington Memorial Hospital
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 91 | 90 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (8.8) | 78.4 (7.8) | 78.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 39 | 88
  Male | 42 | 51 | 93
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 23 | 14 | 37
  Caucasian | 52 | 57 | 109
  Latino | 7 | 9 | 16
  Native American | 1 | 1 | 2
  Asian/Pacific Islander | 4 | 2 | 6
  Other | 3 | 6 | 9
  Declined to provide response | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 91 | 90 | 181
Marital status [Number; unit: participants]
  Married | 35 | 45 | 80
  Single | 11 | 16 | 27
  Divorced | 10 | 7 | 17
  Widowed | 35 | 19 | 54
  Declined to provide response | 0 | 3 | 3
Current living situation [Number; unit: participants]
  Own house/apartment | 82 | 78 | 160
  Living in family member's home | 7 | 6 | 13
  Other | 2 | 3 | 5
  Declined to provide response | 0 | 3 | 3
Who do you live with? [Number; unit: participants]
  Alone | 35 | 20 | 55
  Spouse/partner | 31 | 43 | 74
  Child | 14 | 13 | 27
  Paid caregiver | 2 | 1 | 3
  Other | 9 | 8 | 17
  Declined to provide response | 0 | 5 | 5
Who is your primary caregiver? [Number; unit: participants]
  No one/self | 43 | 33 | 76
  Spouse | 19 | 24 | 43
  Significant other | 0 | 4 | 4
  Child | 11 | 11 | 22
  Paid caregiver | 9 | 6 | 15
  Other | 9 | 8 | 17
  Declined to provide response | 0 | 4 | 4
Current annual income [Number; unit: participants]
  Under $10,000 | 15 | 9 | 24
  $10,000-$19,000 | 9 | 10 | 19
  $20,000-$29,000 | 9 | 5 | 14
  $30,000-$39,000 | 3 | 1 | 4
  $40,000-$49,000 | 0 | 1 | 1
  $50,000 or more | 11 | 11 | 22
  Refused to respond | 44 | 53 | 97
Highest grade completed in school [Number; unit: participants]
  8th grade or less | 1 | 5 | 6
  9th-11th grade | 4 | 5 | 9
  High school graduate | 17 | 13 | 30
  Some college | 27 | 20 | 47
  College graduate | 17 | 19 | 36
  Graduate degree | 10 | 14 | 24
  Doctoral degree | 7 | 4 | 11
  Declined to provide response | 8 | 10 | 18
Chronic condition inventory [Number; unit: participants] — Measure NOT mutually exclusive. Inventory of conditions
  participants
    Cancer | 24 | 20 | 44
    Cardiac disease | 58 | 55 | 113
    Dementia/Alzheimer's disease | 3 | 4 | 7
    Depression | 14 | 32 | 46
    Diabetes | 18 | 23 | 41
    Hypertension | 57 | 54 | 111
    Respiratory disease | 30 | 29 | 59
    Stroke | 7 | 10 | 17
Patient Health Questionnaire 9-item (PHQ-9) [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire, 9-item uses nine questions to asses for depression and has been widely and successfully used in health care research since the early 1990's, particularly in investigations among older adults aged 65 years or more.
  A total score is reported at the end of the questionnaire and scores can range from 0-27 with a higher value indicating more severe or worse depression. Total scores correspond to the following: 0 no depression, 1-4 minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderate severe depression, and 20-27 severe depression.
  units on a scale | 4.33 (3.9) | 6.15 (5.1) | 5.24 (4.5)
Pain (Number Rating Scale) [Mean (Standard Deviation); unit: units on a scale] — The Number Rating Scale is a self-reported measure for pain level that is widely used in US hospitals. Patients are asked to rate their level of pain felt over the last 24-hours on a scale ranging from 0-10, where zero indicates no pain, and 10 is the worst pain imaginable.
  units on a scale | 3.54 (3.4) | 9.18 (1.1) | 6.36 (2.25)
Physical Functioning Index (abbreviated Short Form-12) [Mean (Standard Deviation); unit: units on a scale] — The Short-Form, 12-item is a survey tool to measure physical health and functional level and an abbreviated version of this tool was used in the present study which constituted eight of the 12-items that focused on physical functioning. Response options ranged from 'not limited at all,' to 'limited a lot' and after assigning numerical values to response options, total scores ranged from 0-16 with a higher score corresponding to greater physical limitations.
  units on a scale | 7.67 (5.12) | 7.18 (5.08) | 7.43 (5.1)
Cognition (SPMSQ score) [Mean (Standard Deviation); unit: units on a scale] — The Short Portable Mental Health Questionnaire (SPMSQ) is widely used tool to screen for cognitive impairment. This questionnaire consists of 10 questions and a total score is derived at the end. Scores can range from 0-10 where a low score indicates high cognitive impairment and a high score indicates higher cognitive functioning. The scale has an established cut-off score of 5 where those scoring 5 or higher are cognitively intact to participate in research, understand the study and associated activities, and provide consent. Those scoring below 5 are deemed ineligible.
  units on a scale | 9.08 (1.2) | 9.18 (1.1) | 9.13 (1.15)
Number of health conditions [Mean (Standard Deviation); unit: health conditions] | 6.35 (4.1) | 5.88 (2.9) | 6.17 (3.5)
Number of daily medications [Mean (Standard Deviation); unit: medications] | 7.61 (3.8) | 8.00 (3.8) | 7.81 (3.8)
Discharged home under self-care [Number; unit: participants]
  Yes | 61 | 67 | 128
  No | 30 | 23 | 53
Had inpatient stay or emergency department visit in previous 6 months [Number; unit: participants]
  Yes | 35 | 32 | 67
  No | 56 | 58 | 114
Has Advance Directive [Number; unit: participants]
  Yes | 50 | 46 | 96
  No | 41 | 44 | 85

OUTCOME MEASURES:

1. Primary Outcome: 30-day Hospital Readmission
Description: The outcome measure is the number of readmissions experienced by participants in the Usual Care and Intervention groups within 30-days of their index discharge.
Time Frame: 30-days post hospitalization
Measure: Number; unit: 30-day hospital readmissions
Groups:
- Usual Care: Usual Care in the present study constitutes usual care that is delivered to older adults transitioning from the hospital to home from Huntington Memorial Hospital.
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 91 | 90
30-day hospital readmissions | 11 | 9

2. Secondary Outcome: 30-day Readmission Among Intervention Participants
Description: The outcome measure is the rate of 30-day readmissions among Intervention group participants that declined to receive the in-home social work intervention versus those Intervention group participants that received the in-home social work intervention.
Time Frame: 30-days
Population: Analysis among Intervention group ONLY for this outcome
Measure: Number; unit: 30-day hospital readmissions
Groups:
- Intervention Group: Received Intervention: Patients randomized to the intervention group and received the intervention. SWIFT home intervention: 1 in-home assessment performed by study social worker, another in-home visit performed if needed. Up to 4 telephone contacts performed by study social worker. A maximum of 6 contacts
- Intervention Group: Opt-outs: Patients randomized to the intervention group that refused the intervention.
Arm/Group | Intervention Group: Received Intervention | Intervention Group: Opt-outs
Number analyzed (Participants) | 63 | 27
30-day hospital readmissions | 4 | 5

ADVERSE EVENTS:
Groups:
- Usual Care: Usual care for the present study constituted the usual course of care provided to older adults transitioning from hospital to home from Huntington Memorial Hospital.
Arm/Group | Usual Care | Intervention
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/90
Other Adverse Events (participants affected / at risk) | 0/91 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No